CLINICAL TRIAL: NCT00469222
Title: Phase I Dose Escalation Trial of Hypofractionated Limited-field External Beam Thoracic Radiotherapy for Limited Stage Small Cell Carcinoma of the Lung
Brief Title: Hypofractionated Radiotherapy for Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LU-11-0072 / 23117
Record Dates: First submitted 2007-05-02; First posted 2007-05-04 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2012-03

CONDITIONS: Lung Neoplasm; Small Cell Carcinoma
Keywords: small cell lung cancer; radiotherapy dose escalation
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Small Cell; Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: hypofractionated external beam

SUMMARY:
Current treatments for limited stage small cell lung cancer have poor cure rates. The addition of chest radiation to chemotherapy improves cure rates, but these cancers still come back in the chest 30-50% of the time. Two factors which can improve control and cure rates for this cancer are increasing the chest radiation dose and minimizing the overall time it takes to complete radiation treatments. One method to achieve both of these goals is to give more radiation each day. This study is meant to study how tolerable and effective it would be to increase the intensity of chest radiation for small cell lung cancer patients by increasing the daily radiation dose. We aim to find the highest dose of chest radiotherapy that can be safely given with chemotherapy using this strategy. Patients in this trial will be monitored before, during and after their radiation and chemotherapy treatments for treatment side-effects, how effective treatments are at controlling their cancer and quality of life changes. Results from this trial will help to define more effective radiotherapy doses which are tolerable for this type of lung cancer and the quality of life changes patients experience when they undergo these treatments.

DETAILED DESCRIPTION:
Local control and overall survival rates associated with the standard chemotherapy and radiotherapy given for limited stage small cell lung cancer are poor and emerging evidence from several studies suggests that intensifying the radiotherapy dose given may further improve patient outcomes, but at the cost of increased radiotherapy side effects. This proposal aims to study a novel method of intensifying chest radiotherapy dose via increasing the daily radiotherapy dose which is directed at regions of visible disease only. This strategy allows for delivery of increased radiation doses without prolonging overall treatment time and allowing potential regrowth of cancer cells. We aim to determine the maximum radiation dose which can be safely given with chemotherapy for limited stage small cell lung cancer and study the effects this type of radiation regimen with chemotherapy has on patient side effects and quality of life. Results from this trial will contribute to the development of the ideal radiotherapy regimen for limited stage small cell lung cancer. Our results will add to the literature studying the effects dose-intense radiation strategies for lung cancer have on patient quality of life.

ELIGIBILITY:
Inclusion Criteria:

* patients with histologically or cytologically proven newly diagnosed small cell lung cancer
* confirmation from the treating radiation oncologist that the patient has limited stage disease (i.e. disease that can be encompassed by radiotherapy portals without exposing patient to excessive risk of radiation lung injury)
* adequate pulmonary function tests (FEV-1 >1.0, DLCO >50%)
* patients of childbearing potential must practice adequate contraception
* age greater than 18 years
* Karnofsky performance status greater than 70
* adequate hematologic, hepatic and renal function: Hb>100g/L, WBC > 4.0x109/L, neutrophils > 1.0x109/L, platelets > 100,000x109/L, calculated GFR based on Cockcroft-Gault formula of >60mL/min (NOTE: for cisplatin, GFR must be above 60ml/min; if less than 60ml/min the patient can not receive cisplatin but could be considered for carboplatin)
* patients must sign a study specific informed consent form

Exclusion Criteria:

* patient who have undergone complete or subtotal tumour resection
* evidence of non-small cell histology
* pericardial or pleural effusion on radiologic investigations regardless of cytology
* patients cannot be treated with 3DCRT with adherence to the dose volume constraints
* prior or concurrent malignancy except non-melanomatous skin cancer unless disease-free for at least 5 years
* prior radiotherapy to the thorax or neck
* prior chemotherapy
* patients with myocardial infarction within the preceding 6 months or symptomatic heart disease, including angina, congestive heart failure, uncontrolled arrhythmias
* compromised lung function with inadequate pulmonary function tests (FEV-1<1.0, DLCO <50%)
* pregnancy (patients with childbearing potential must practice appropriate contraception)
* patients who have not had the pre-treatment evaluations outlined in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Rates of acute grade 3 or higher radiotherapy toxicities

SECONDARY OUTCOMES:
Overall survival and disease free survival, patient related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Don Yee, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada